CLINICAL TRIAL: NCT03742297
Title: Induction Therapy With Bortezomib-melphalan and Prednisone (VMP) Followed by Lenalidomide and Dexamethasone (Rd) Versus Carfilzomib, Lenalidomide and Dexamethasone (KRd) Plus/Minus Daratumumab, 18 Cycles, Followed by Consolidation and Maintenance Therapy With Lenalidomide and Daratumumab: Phase III, Multicenter, Randomized Trial for Elderly Fit Newly Diagnosed Multiple Myeloma Patients Aged Between 65 and 80 Years
Brief Title: Treatment for Elderly Fit Newly Diagnosed Multiple Myeloma Patients Aged Between 65 and 80 Years
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM2017FIT
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Newly Diagnosed Multiple Myeloma
MeSH Terms: interventions — Lenalidomide; carfilzomib; Bortezomib; daratumumab; Dexamethasone; Prednisone; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VMP x 9 + Lenalidomida-dexamethasone x 9 (Active Comparator): Bortezomib-melfalán-prednisone. Melfalán: 9mg/m2D1-4. Prednisone: 60mg/m2D1-4. Bortezomib: 1.3mg/m2 One 6 week cycleD1, 4, 8, 11, 22, 25, 29 and 32; followed by eight4-week cycleD1, 8, 15 and 22 Lenalidomida-dexametasona at low dose
  Interventions: Drug: Lenalidomide.; Drug: Bortezomib; Drug: Dexamethasone; Drug: Prednisone; Drug: Melphalan
- Carfilzomib-lenalidomida-dexamethasone regimen (Experimental): carfilzomib: 1 st cycle: 20mg/m2 day 1 and 36 mg/m2 days 2, 8, 9 & 15, 16. 2nd cycle: 36 mg/m2 days 1, 2, 8, 9 & 15, 16. Cycles 3-18: 56 mg/m2 days 1, 8 & 15.Lenalidomida: 25 mg, d1-21 Dexamethasone : 40 mg, d1, 8, 15, 2218 28-day cycle
  Interventions: Drug: Lenalidomide.; Drug: Carfilzomib; Drug: Dexamethasone
- Carfilzomib-lenalidomida-dexamethason with daratumumab (Experimental): Carfilzomib: 1 st cycle: 20mg/m2 day 1 and 36 mg/m2 days 2, 8, 9 & 15, 16. 2nd cycle: 36 mg/m2 days 1, 2, 8, 9 & 15, 16. Cycles 3-18: 56 mg/m2 days 1, 8 & 15. Lenalidomida: 25 mg, d1-21 Dexamethasone: 40 mg, d1, 8, 15, 22. Daratumumab 1800mg SC Days 1, 8, 15, 22 of cycles 1-2; Days 1 and 15 of cycles 3 and 4; Day 1 of cycles 5 to 18
  Interventions: Drug: Lenalidomide.; Drug: Carfilzomib; Drug: Daratumumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide. — Lenalidomide
Drug: Carfilzomib — Carfilzomib
  Arms: Carfilzomib-lenalidomida-dexamethason with daratumumab; Carfilzomib-lenalidomida-dexamethasone regimen
Drug: Bortezomib — Bortezomib
  Arms: VMP x 9 + Lenalidomida-dexamethasone x 9
Drug: Daratumumab — Daratumumab
  Arms: Carfilzomib-lenalidomida-dexamethason with daratumumab
Drug: Dexamethasone — Dexamethasone
Drug: Prednisone — Prednisone
  Arms: VMP x 9 + Lenalidomida-dexamethasone x 9
Drug: Melphalan — Melphalan
  Arms: VMP x 9 + Lenalidomida-dexamethasone x 9

SUMMARY:
The study is designed as a randomized, controlled, open-label, assessor blind, multicenter superiority trial with three parallel groups, and primary endpoint of immunophenotypic complete responses at 18 months after randomization. Block randomization will be performed with a 1:1:1 allocation ratio.

Patients will be randomized up front to 3 arms. Patients will receive "standard" PETHEMA arm for fit elderly VMP x 9 + Rd x 9 (arm 1, control arm), a KRd regimen (arm 2a) (18 cycles) or a Carfilzomib-lenalidomida-dexametasona regimen combined with DARATUMUMAB (arm 2b) (18 cycles).

DETAILED DESCRIPTION:
After 18 cycles, patients not having received daratumumab before (arm 1 and 2a), will receive consolidation with 4 cycles of Lenalidomida-dexamethasone at low dose-DARATUMUMAB.

At this point (after 22 months on treatment for the VMP-Rd and KRd arm and after 18 months of the Carfilzomib-lenalidomida-dexametasona-DARATUMUMAB arm) patients will be stratified according MRD status by flow and in both MRD- and MRD+ groups, patients will be randomized with a 1:1 allocation ratio to:

1. no further treatment or
2. continuous treatment with DARATUMUMAB-R (daratumumab plus lenalidomide up to 2 years and then lenalidomide continuous until progression).

Patients on no maintenance that show biological relapse will be rechallenged with DARATUMUMAB-R.

The translational part will be very robust with dysplasia monitoring (especially relevant for the Bortezomib-melfalán-prednisona + Lenalidomida-dexamethasone at low dose arm), clonal evolution/resistance follow up and immune reconstitution longitudinal follow up alongside with MRD status (at diagnosis, 9 months, 18 months, 22 months and treatment discontinuation).

The trial is designed as a two-stage study (induction, followed by consolidation and maintenance). The first stage is confirmatory and addresses the primary efficacy objective. The second stage is exploratory and addresses the secondary efficacy and safety objectives.

In the first stage, investigators will compare an optimized standard induction Bortezomib, talidomida and prednisone followed by Rd (18 cycles) versus KRd, that will be tested in this trial with or without daratumumab x 18 cycles. The main objective in this stage will be to compare the immunophenotypic complete response rate assessed by next generation flow at the end of induction.

The second stage is exploratory and includes the consolidation and maintenance phases. In this second stage, the main objectives are:

1. To compare the above mentioned induction strategies in terms of PFS at the end of the different treatment phases (induction, consolidation and maintenance).
2. To investigate the capacity of consolidation with daratumumab-lenalidomide to reduce MRD levels in patients treated in the control arm as well as those that received KRd without daratumumab. In addition we will explore if this short consolidation can abrogate the potential benefit of a prolonged induction with KRd+daratumumab
3. To explore the value of maintenance therapy according to MRD status (positive or negative) to prolong PFS (after a second randomization to receive or not maintenance therapy with lenalidomide and daratumumab) In order to prevent a potential treatment deficiency for patients randomized to "no-maintenance" in both MRD+ and MRD- subgroups, they will be offered to be re-challenged with lenalidomide-daratumumab as soon as they have a biological progression and have been censored for PFS. Moreover, if 30% of the patients randomized to "no-maintenance" relapse or progress during the first year, the protocol will be amended so that all patients receive maintenance therapy.

Investigators consider that the here proposed multidrug sequential "intensive" approach designed to obtain the best possible and most durable response, assessed through the kinetics of MRD clearance, may have an impact in establishing future clinical practice in fit elderly patients. Moreover, in addition to the MRD analysis (based on next generation flow (NGF), NGS and CT-PET) comprehensive biological investigations, including immunoprofile, clonal selection, analysis of dysplastic features and circulating tumor cells, are planned in order to better understand the relationship between patients outcome and myeloma biology.

The overall treatment plan has been designed for NDMM patients not candidates to SCT strategies but fit enough to tolerate a relatively intensive therapeutic strategy. According to the International Myeloma Working Group guidelines as well as the results obtained in our GEM2010 trial for elderly patients, we have decided to restrict this trial to fit elderly patients aged between 65 and 80 years because in our experience patients older than 80 years usually intensive treatments are poorly tolerated [1].

Investigators will evaluate the frailty using a comprehensive health status assessment scale (Geriatric Assessment in Hematology, GAH scale, annex 11), already validated in patients with hematological diseases and preliminary results in multiple myeloma patients

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed multiple myeloma patients who require start active treatment according to the IMWG published in 2014
* Age between 65 and 80 years, both included
* Fit patient assessed using the comprehensive health status assessment scale (Geriatric Assessment in Hematology, GAH scale, annex 11) (0-94 points GAH scale). Patients with a punctuation ≤42 will be included.
* Signed informed consent
* Patients must have measurable disease, defined as follows:

For secretory Multiple Myeloma, measurable disease is defined as the presence of quantifiable monoclonal component, ≥ 0.5 g/dL or, the urine light chains excretion is 200 mg/24h or higher.

For poor secretory or non secretory Multiple Myeloma, the level of the affected serum free light chain must be ≥ 10 mg/dL (≥ 100 mg/L, with an abnormal free light-chain ratio)

* Eastern Cooperative Oncology Group (ECOG) Performance status ≤2
* Life expectancy more than 3 months
* Adequate organ functions:

Platelet count ≥ 50000/mm3, hemoglobin ≥ 8 g/dl and absolute neutrophil count ≥ 1000/mm3. Lower values are allowed only if they are due to BM infiltration.

Aspartate Transaminase (AST) and Alanine Transaminase (ALT) ≤ 2.5 x Upper Limit of Normal.

Total bilirubin: ≤2 x Upper Limit of Normal. Serum creatinine ≤ 2 mg/dl. Calcium ≤14mg/dl or corrected serum calcium ≤14mg/dl in patients whose albumin level is out of range Left ventricle ejection fraction ≥ 40%

* At the discretion of the investigator patient must be able to adhere to all study requirements.
* Male patients that receives lenalidomide should commit to use of a condom while taking the study drug every time he has sexual contact with a pregnant female of female of childbearing potential even if he has undergone a successful vasectomy; or practice complete abstinence (when this is the preferred and usual lifestyle of the subject); including during periods of dose interruptions and for at least 30 days after treatment completion. Also males under lenalidomide should commit not to donate semen or sperm during study drug treatment, including during periods of dose interruptions, and for at least 90 days after treatment completion.

NOTE: Given the age of patients to be included on this Clinical Trial (between 65 and 80 years, both included), there is no possibility of Females of Childbearing Potential (FCBP), therefore the Pregnancy Prevention Program (annex 12) has been modified accordingly.

Exclusion Criteria:

* Patients older than 81 years or younger than 65
* Patients that do not qualify for fit according to the GAH scale (annex 11) (>43 points GAH scale)
* Patients who have previously received treatment for multiple myeloma, except for steroid pulses in case of emergency, the administration of bisphosphonates or antialgesic radiotherapy or due to the presence of plasmacytomas requiring some emergency.
* Men who does not agree to use a condom every time he has sexual contact with a pregnant female or female of childbearing potential, even if he has undergone a successful vasectomy, or men who does not agree to practice complete abstinence (if this is the preferred and usual lifestyle of the subject).
* Left ventricular ejection fraction <40% Prior history of malignancies, other than multiple myeloma (except for basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or the breast), unless the patient has been free of the disease for ≥ 5 years.
* Other relevant diseases or adverse clinical conditions:

Myocardial infarction within the 6 months prior to inclusion in the clinical trial A NYHA functional class III-IV, heart failure, uncontrolled angina, uncontrolled ventricular arrhythmia or acute ischemia detected electrocardiographically or conduction system anomalies.

History of significant neurological or psychiatric disorders. Active infection. Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).

Poorly controlled arterial hypertension. Any serious medical condition or psychiatric illness that would interfere in understanding of the informed consent form.

* Human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive or active hepatitis C infection
* Limitation of the patient's ability to comply with the treatment or follow-up protocol.
* Uncontrolled endocrine diseases (i.e. diabetes mellitus, hypothyroidism or hyperthyroidism) (i.e. requiring relevant changes in medication within the last month, or hospital admission within the last 3 months).
* Patients having a peripheral neuropathy ≥ Grade 2 within the 14 days prior to inclusion.
* Known hypersensibility to any of the study drugs or their excipients.
* Patients treated with any investigational drug during the previous 30 days.
* Patients with acute diffuse infiltrative pulmonary disease and/or pericardial disease.
* Patients who are unable or unwilling to undergo antithrombotic therapy.
* Patients with severe chronic obstructive pulmonary disease (COPD) or asthma with forced expiratory volume in the first minute (FEVI) less than 50%.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 462 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy in terms of numbers of compleat responses | 18 months
  Rate of immunophenotypic complete responses at 18 months, of the standard treatment in Spain for newly diagnosed multiple myeloma patients not candidates to stem cell transplantation,

CONTACTS AND LOCATIONS:
Overall Officials: Jesús F San Miguel, Study Chair — Clínica Universidad de Navarra; Joan Blade, Dr, Study Chair — Hospital Clinic of Barcelona; Juan Jose Lahuerta, Dr, Study Chair — Hospital 12 de Octubre
Locations (58):
- Spain (58):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Germans Trias i Pujol (ICO Badalona), Badalona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - ICO L´Hospitalet, Barcelona
  - Hospital Universitario de Cruces, Bilbao
  - Complejo Hospitalario de Cáceres, Cáceres
  - Complejo Hospitalario Regional Reina Sofía, Córdoba
  - Hospital de Cabueñes, Gijón
  - Hospital Universitari Dr. Josep Trueta (ICO Girona), Girona
  - Hospital de Especialidades de Jerez de la Frontera, Jerez de la Frontera
  - Complejo Hospitalario Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital San Pedro, Logroño
  - Complejo Hospitalario Lucus Augusti, Lugo
  - Hospital 12 de octubre, Madrid
  - Hospital clínico San Carlos, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - HU Gregorio Marañón, Madrid
  - Hospital San Joan de Deu (Althaia), Manresa
  - Hospital Costa del Sol, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital General Universitario Santa Lucía, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Clinica Universitaria de Navarra, Pamplona
  - Complejo Hospitalario de Navarra, Pamplona
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Donostia, San Sebastián
  - Complejo Hospitalario Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - H. Universitario Virgen de Rocío, Seville
  - Hospital Nuestra Señona de Valme, Seville
  - Hospital Universitari Joan XXIII de Tarragona, Tarragona
  - Complejo Hospitalario de Toledo (Virgen de la Salud), Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic la Fe, Valencia
  - Hospital Universitario Dr. Peset Aleixandre, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital Clínico Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mateos MV, Paiva B, Cedena MT, Puig N, Sureda-Balari AM, de la Calle VG, Oriol A, Ocio EM, Rosinol L, Montes YG, Bargay J, Garcia MEG, Lakhwani S, Payer AR, Suarez-Cabrera A, Blanchard MJ, Garzon S, Montero FC, Cabanas V, de Oteyza JP, Gironella M, Martinez-Lopez J, Casasus AIT, Delgado-Beltran MP, Prieto E, Lahuerta JJ, Blade J, San-Miguel J. Induction therapy with bortezomib, melphalan, and prednisone followed by lenalidomide and dexamethasone versus carfilzomib, lenalidomide, and dexamethasone with or without daratumumab in older, fit patients with newly diagnosed multiple myeloma (GEM-2017FIT): a phase 3, open-label, multicentre, randomised clinical trial. Lancet Haematol. 2025 Aug;12(8):e588-e598. doi: 10.1016/S2352-3026(25)00143-7. PMID 40769684